CLINICAL TRIAL: NCT02163915
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Multiple Rising Doses of TAK-137 in Adult Subjects With Attention-Deficit/Hyperactivity Disorder
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Doses of TAK-137 in Adults With Attention-Deficit/Hyperactivity Disorder.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To allow evaluation of emerging non-clinical data (see detailed description below)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-137_102; U1111-1152-6846 (Other: World Health Organization)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: Drug therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — TAK-137

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: TAK-137 0.5 mg (Experimental): TAK-137 0.5 mg, tablets, orally once on Days 1-7.
  Interventions: Drug: TAK-137
- Cohort 2: TAK-137 2 mg (Experimental): TAK-137 2 mg, tablets, orally once on Days 1-7.
  Interventions: Drug: TAK-137
- Cohort 3: TAK-137 5 mg (Experimental): TAK-137 5 mg, tablets, orally once on Days 1-7.
  Interventions: Drug: TAK-137
- Cohort 4: TAK-137 10 mg (Experimental): TAK-137 10 mg, tablets, orally once on Days 1-7.
  Interventions: Drug: TAK-137
- Cohort 5: TAK-137 TBD (Experimental): TAK-137, tablets, orally once on Days 1-7. Dose to be determined from data collected in Cohorts 1-3.
  Interventions: Drug: TAK-137
- Cohorts 1-5: Placebo (Experimental): TAK-137 placebo-matching tablets, orally, once on Days 1-7.
  Interventions: Drug: TAK-137 Placebo

INTERVENTIONS:
Drug: TAK-137 — TAK-137 tablets
  Arms: Cohort 1: TAK-137 0.5 mg; Cohort 2: TAK-137 2 mg; Cohort 3: TAK-137 5 mg; Cohort 4: TAK-137 10 mg; Cohort 5: TAK-137 TBD
Drug: TAK-137 Placebo — TAK-137 placebo-matching tablets
  Arms: Cohorts 1-5: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of TAK-137 when administered as multiple oral doses in adults with attention-deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-137. TAK-137 is being tested to find a safe and well-tolerated dose and to assess how TAK-137 is metabolized in people with attention-deficit/ hyperactivity disorder (ADHD). This study will look at side effects and lab results in people who take TAK-137. This study is designed as a randomized, sequential-cohort, multiple rising dose study.

Therefore, the TAK-137 2 mg Cohort will not start until the TAK-137 0.5 mg Cohort has completed, etc.

This trial will be conducted in the United States. The overall time to participate in this study is up to 42 days. Participants will make at least 2 visits to the clinic, including one 9-day period of confinement to the clinic. All participants will be contacted by telephone 7 days after the last dose of study drug for a follow-up assessment.

A decision was made to terminate this study so that emerging data from preclinical studies could be further assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female adult who is 18 to 55 years of age, inclusive.
2. Weighs at least 45 kg and has a body mass index (BMI) between 18 and 30.0 kg/m^2, inclusive at Screening.
3. Has a documented diagnosis of attention-deficit/hyperactivity disorder (ADHD) for a minimum of 1 year.
4. Is willing to discontinue all medications to treat adult ADHD (eg, stimulants, antidepressants) and all other medications and dietary products as specified in the protocol, from Day -7 until Follow-up phone call (Day 14).

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has uncontrolled, clinically significant neurologic (including mildly abnormal or significantly abnormal EEG at screening), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder (other than ADHD), or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
3. Has previously had a seizure or convulsion (lifetime), including absence seizure and febrile convulsion.
4. Has a positive urine drug result for drugs of abuse other than amphetamines or other medications to treat ADHD or positive result for alcohol at Screening or Check-in (Day -1).
5. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products.
6. Is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during such time period.
7. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Marlton, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 23 May 2014 to 03 November 2014.
Pre-assignment Details: Participants with a historical diagnosis of attention-deficit/hyperactivity disorder (ADHD) were enrolled in one of the five cohorts to receive TAK-137 (0.5 milligram [mg], 2 mg, 5 mg, 10 mg, or matching placebo) once daily for up to 7 days.
Groups:
- Cohorts 1-4: Placebo: TAK-137 placebo-matching tablets, orally, once on Days 1-7 under fasting conditions.
- Cohort 1: TAK-137 0.5 mg: TAK-137 0.5 mg, tablets, orally once on Days 1-7 under fasting condition.
- Cohort 2: TAK-137 2 mg: TAK-137 2 mg, tablets, orally once on Days 1-7 under fasting condition.
- Cohort 3: TAK-137 5 mg: TAK-137 5 mg, tablets, orally once on Days 1-7 under fasting condition.
- Cohort 4: TAK-137 10 mg: TAK-137 10 mg, tablets, orally once on Days 1-7 under fasting condition.
Period: Overall Study
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Started | 10 | 8 | 10 | 9 | 10
Completed | 7 | 8 | 8 | 6 | 6
Not Completed | 3 | 0 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 2 | 2
Not completed — Study termination | 1 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg | Total
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (10.59) | 33.0 (9.65) | 28.6 (8.75) | 32.6 (10.73) | 31.6 (11.68) | 30.6 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 2 | 3 | 12
  Male | 5 | 7 | 9 | 7 | 7 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5 | 2 | 6 | 4 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  White | 4 | 3 | 4 | 5 | 3 | 19
  Multiracial | 1 | 2 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 2 | 1 | 3 | 8
  Non-Hispanic or Latino | 8 | 8 | 8 | 8 | 7 | 39
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.8 (7.96) | 172.4 (9.07) | 171.7 (7.09) | 174.8 (7.36) | 172.4 (5.23) | 172.6 (7.13)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.42 (10.211) | 76.01 (14.537) | 75.11 (14.376) | 79.61 (9.205) | 74.73 (13.815) | 76.54 (12.777)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.25 (3.182) | 25.46 (3.408) | 25.36 (3.942) | 26.02 (2.204) | 25.09 (3.969) | 25.64 (3.303)
Caffeine Consumption [Number; unit: participants]
  Had caffeine consumption | 7 | 5 | 6 | 7 | 4 | 29
  Had no caffeine consumption | 3 | 3 | 4 | 2 | 6 | 18
Smoking Status [Number; unit: participants] — The baseline characteristic was categorized as never smoked, current smoker and ex-smoker. There were no participants available under current smoker.
  participants
    Never smoked | 8 | 7 | 8 | 8 | 9 | 40
    Ex-smoker | 2 | 1 | 2 | 1 | 1 | 7
Alcohol consumption [Number; unit: participants]
  Never drank | 5 | 4 | 5 | 4 | 9 | 27
  Current drinker | 4 | 3 | 5 | 4 | 1 | 17
  Ex-drinker | 1 | 1 | 0 | 1 | 0 | 3
Female Reproductive Status [Number; unit: participants] — The baseline measure was categorized as Surgically sterile: permanent method of contraception; Female of childbearing potential; and Not applicable: participant was male.
  participants
    Surgically sterile | 1 | 1 | 0 | 1 | 0 | 3
    Female of childbearing potential | 4 | 0 | 1 | 1 | 3 | 9
    Not applicable | 5 | 7 | 9 | 7 | 7 | 35
ADHD Category [Number; unit: participants] — As per national institute of mental health (NIMH) ADHA was categorized as Combined: participants who had greater than equal to (>=) 6 symptoms of inattention and hyperactivity-impulsivity; Hyperactive/impulsive: participants who had >=6 symptoms of hyperactivity-impulsivity and less than (<) 6 symptoms of inattention; and Inattentive; participants who had >=6 symptoms of inattention and <6 symptoms of hyperactivity-impulsivity. There were no participants available under hyperactive/impulsive.
  participants
    Combined | 9 | 8 | 8 | 9 | 9 | 43
    Inattentive | 1 | 0 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 up to Day 14
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10
percentage of participants | 50.0 | 62.5 | 0 | 66.7 | 20.0

2. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Time Frame: Day 1 up to Day 8
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10
percentage of participants | 0 | 12.5 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Pulse Measurements at Least Once Post Dose
Time Frame: Day 1 up to Day 8
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10
percentage of participants
  Supine, After 5 Minutes: < 50 bpm | 50 | 37.5 | 50 | 22.2 | 40
  Standing, After 1 Minute: < 50 bpm | 10 | 0 | 0 | 11.1 | 0
  Standing, After 1 Minute: > 120 bpm | 10 | 0 | 10 | 0 | 40
  Standing, After 3 Minutes: < 50 bpm | 20 | 12.5 | 20 | 22.2 | 0
  Standing, After 3 Minutes: > 120 bpm | 30 | 0 | 10 | 0 | 50

4. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Blood Pressure Measurements at Least Once Post Dose
Time Frame: Day 1 up to Day 8
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10
percentage of participants
  SBP: Supine, After 5 Minutes: < 85 mmHg | 10 | 0 | 0 | 11.1 | 10
  SBP: Standing, After 3 Minutes: <85 mmHg | 0 | 0 | 0 | 0 | 10
  DBP: Supine, After 5 Minutes: <50 mmHg | 30 | 25 | 10 | 44.4 | 0
  DBP: Standing, After 1 Minute: <50 mmHg | 30 | 0 | 10 | 22.2 | 0
  DBP: Standing, After 1 Minute: >110 mmHg | 0 | 0 | 0 | 0 | 10
  DBP: Standing, After 3 Minutes: <50 mmHg | 30 | 25 | 30 | 44.4 | 20
  DBP: Standing, After 3 Minutes: >110 mmHg | 0 | 0 | 0 | 11.1 | 10

5. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Heart Rate Measurements at Least Once Post Dose
Time Frame: Day 1 up to Day 8
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10
percentage of participants | 30 | 25 | 30 | 22.2 | 30

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-137
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: Pharmacokinetic analysis set was defined as all participants who received at least one dose of study drug and had at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 8 | 10 | 8 | 10
nanogram per milliliter (ng/mL) | 8.32 (2.651) | 28.04 (7.554) | 64.91 (24.592) | 103.13 (27.822)

7. Secondary Outcome: Cmax, ss: Maximum Observed Plasma Concentration at Steady State for TAK-137
Description: Maximum observed steady-state plasma concentration during a dosing interval.
Time Frame: Day 7 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 8 | 8 | 6 | 6
ng/mL | 7.79 (2.039) | 38.01 (22.749) | 86.25 (35.079) | 176.25 (113.096)

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-137
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Days 1 and 7 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 8 | 10 | 8 | 10
hours
  Day 1 (n= 8, 10, 8, 10) | 1.560 (2.039) [1.00 to 3.02] | 1.750 (22.749) [1.00 to 4.00] | 2.060 (35.079) [1.50 to 4.02] | 4.000 (113.096) [1.00 to 4.05]
  Day 7 (n= 8, 8, 6, 6) | 1.015 [1.00 to 2.00] | 1.750 [1.00 to 4.00] | 3.500 [2.00 to 4.00] | 2.000 [1.00 to 3.00]

9. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-137
Description: Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval.
Time Frame: Days 1 and 7 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 8 | 10 | 8 | 10
nanogram hours per milliliter (ng*hr/mL)
  Day 1 (n= 8, 10, 8, 10) | 73.5 (37.87) [1.00 to 3.02] | 265.3 (156.89) [1.00 to 4.00] | 717.1 (432.37) [1.50 to 4.02] | 1442.8 (621.57) [1.00 to 4.05]
  Day 7 (n= 8, 8, 6, 4) | 52.9 (24.15) [1.00 to 2.00] | 438.4 (600.42) [1.00 to 4.00] | 1224.0 (689.80) [2.00 to 4.00] | 3288.5 (3189.13) [1.00 to 3.00]

10. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: Day 1 up to Day 8
Population: Safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Number analyzed (Participants) | 10 | 8 | 10 | 9 | 10
percentage of participants
  PR Interval: ≤80 msec | 0 | 0 | 10 | 0 | 0
  PR Interval: ≥200 msec | 0 | 25 | 30 | 22.2 | 10
  QRS Interval: ≤80 msec | 10 | 0 | 20 | 22.2 | 20
  QT Interval: ≥460 msec | 0 | 0 | 10 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug (Day 7).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohorts 1-4: Placebo | Cohort 1: TAK-137 0.5 mg | Cohort 2: TAK-137 2 mg | Cohort 3: TAK-137 5 mg | Cohort 4: TAK-137 10 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 5/8 | 0/10 | 6/9 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-4: Placebo (N=10) | Cohort 1: TAK-137 0.5 mg (N=8) | Cohort 2: TAK-137 2 mg (N=10) | Cohort 3: TAK-137 5 mg (N=9) | Cohort 4: TAK-137 10 mg (N=10)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Electroencephalogram abnormal (Investigations) | 0 | 3 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Infusion site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.